CLINICAL TRIAL: NCT01648192
Title: A Phase I, Randomized, Single-Blind, Three-Period Cross-Over, Placebo-Controlled, Single Oral Dose, Dose-Escalation (Part 1), Fixed Sequence, and Repeat Dose (Part 2) Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of Losmapimod in Healthy Japanese Subjects.
Brief Title: Phase I Study of GW856553 (Losmapimod)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 116681
Record Dates: First submitted 2012-07-12; First posted 2012-07-24 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- 2.5 mg (Experimental): Losmapimod for single dose
  Interventions: Drug: Losmapimod for single dose
- 7.5 mg (Experimental): Losmapimod for single dose
  Interventions: Drug: Losmapimod for single dose
- 20 mg (Experimental): Losmapimod for single dose
  Interventions: Drug: Losmapimod for single dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Losmapimod for single dose
- 7.5 mg BID (Experimental): Losmapimod for repeat dose (14 days)
  Interventions: Drug: Losmapimod for repeat dose
- Placebo BID (Placebo Comparator): Placebo
  Interventions: Drug: Losmapimod for repeat dose

INTERVENTIONS:
Drug: Losmapimod for single dose — Film coated white tablet
  Arms: 2.5 mg; 20 mg; 7.5 mg; Placebo
Drug: Losmapimod for repeat dose — Film coated white tablet
  Arms: 7.5 mg BID; Placebo BID

SUMMARY:
This study is the first study of losmapimod in Japanese subjects. This study will be a single-center, single blind, phase I and two part study to characterize the safety, tolerability, pharmacokinetic and pharmacodynamic profiles in healthy Japanese volunteers (male and female of non-childbearing potential). Part1 will be a single dose, randomized, three-period, placebo-controlled and dose escalation part. Each subject will participate in 3 dosing sessions, and receive, on separate days, three of four treatments of losmapimod 2.5, 7.5 and 20 mg, and the matching placebo in the fasted state after overnight fast (at least 10 hours). The design incorporates sufficient washout between treatments (at least 7 days after the previous administration), and is an efficient design for the study objectives. Part 2 will be a fixed dose and placebo-controlled part. Each subject will participate in one dosing session, and receive losmapimod 7.5 mg or the matching placebo twice daily in the fasted state for 14 days. Only subjects will be blind to the sequence and dose studied. The study will include the placebo treatment to allow a valid evaluation of adverse events attributable to treatment versus those independent of treatment. Approximately 18 subjects in each part will receive treatments of losmapimod and/or placebo in the design. The primary objective of the study is to characterize the safety and tolerability of single doses and repeat doses of losmapimod in healthy Japanese subjects. Serial pharmacokinetic samples will be collected and safety assessments will be performed following each dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Male or female between 20 and 55 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods. This criterion must be followed from the time of the first dose of study medication until follow-up visit.
* Body weight >= 45 kg and BMI within the range 18.5 - 29.0 kg/m2 (inclusive).
* Japanese defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. Japanese subjects must not have lived outside of Japan for more than 10 years.
* ALT, alkaline phosphatase and bilirubin <= 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Single QTc, QTcB or QTcF < 450 msec.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of greater than 21 units for men and 14 for women or an average daily intake of greater than 3 units. One unit is equivalent to a 285 mL glass of full strength beer or 425 mL schooner of light beer or 1 (30 mL) measure of spirits or 1 glass (100 mL) of wine (NHMRC Guidelines [NHMRC, 2009])
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Pregnant females as determined by positive urine hCG test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2012-10-26 (Actual); Study Completion 2012-10-26 (Actual)

PRIMARY OUTCOMES:
Adverse events | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Number of participants with adverse events as a measure of safety and tolerability (evaluated by the result of Clinical safety laboratory tests, vital signs and 12-lead ECG).
AUC(0-t) | up to 96h post dose.
  Area under the concentration-time curve from pre-dose to last time of quantifiable concentration of losmapimod and GSK198602 (inactive metabolite) (Single dose only).
AUC(0-inf) | up to 96h post dose.
  Area under the concentration-time curve from time pre-dose extrapolated to infinite time of losmapimod and GSK198602 (Single dose only).
AUC(0-tau) | up to 17 days post dose.
  Area under the concentration-time curve over the dosing interval of losmapimod and GSK198602 (Repeat dose only).
Cmax | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Maximum observed concentration of losmapimod and GSK198602.
tmax | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Time of occurrence of Cmax of losmapimod and GSK198602.
t1/2 | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Terminal phase half-life of losmapimod and GSK198602
accumulation ratios | up to 17 days post dose.
  accumulation ratios of losmapimod and GSK198602 (Repeat dose only).

SECONDARY OUTCOMES:
hsCRP | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Change from baseline in hsCRP after the oral dose of losmapimod.
phosphorylated HSP27 | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Change from baseline in phosphorylated HSP27 assayed following ex vivo stimulation of cells in wholeblood.
%AUCex | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Percentage of AUC(0-inf) obtained by extrapolation of losmapimod and GSK198602.
tlast | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Time of last quantifiable concentration of losmapimod and GSK198602.
λz | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Terminal phase rate constant of losmapimod and GSK198602.
CL/F | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Apparent clearance following oral dosing of losmapimod.
Vz/F | Single dose: up to 96h post dose. Repeat dose: up to 17 days post dose.
  Apparent volume of distribution following oral dosing of losmapimod.
AUC(0-inf) | up to 17 days post dose.
  Area under the concentration-time curve from time pre-dose extrapolated to infinite time of losmapimod and GSK198602 (Repeat dose only).

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 116681 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/116681?search=study&search_terms=116681#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 116681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 116681 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register